CLINICAL TRIAL: NCT05312242
Title: Introduction of Multiple Micronutrient Supplementation to Antenatal Care in Bamako, Mali
Brief Title: Introduction of MMS to Antenatal Care in Bamako, Mali
Acronym: MAMAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Jhpiego (Other); Bill and Melinda Gates Foundation (Other); Center for Vaccine Development - Mali (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00017475
Record Dates: First submitted 2022-01-27; First posted 2022-04-05 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-02

CONDITIONS: Adherence, Medication
Keywords: Multiple Micronutrient Supplements (MMS); Adherence; Acceptability; Implementation Research; Antenatal Care
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: To examine differences in acceptability and adherence across three different approaches to antenatal micronutrient supplementation within the context of ANC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IFA + Standard of Care (Active Comparator): Iron and Folic Acid (IFA) tablets dispensed 30 tablets at a time + standard of care [Represents standard of care comparison]
  Interventions: Dietary Supplement: Iron Folic Acid Supplement
- MMS 30 + novel counseling (Experimental): MMS dispensed 30 tablets at a time (MMS 30) with novel counseling
  Interventions: Dietary Supplement: United Nations International Multiple Micronutrient Antenatal Preparation (UNIMMAP) MMS
- MMS 180 + novel counseling (Experimental): MMS dispensed 180 tablets at a time (MMS 30) with novel counseling
  Interventions: Dietary Supplement: United Nations International Multiple Micronutrient Antenatal Preparation (UNIMMAP) MMS

INTERVENTIONS:
Dietary Supplement: United Nations International Multiple Micronutrient Antenatal Preparation (UNIMMAP) MMS — Introduction of UNIMMAP MMS along with novel counseling strategies to increase acceptability and adherence to prenatal supplementation
  Other Names: novel counseling strategies
  Arms: MMS 180 + novel counseling; MMS 30 + novel counseling
Dietary Supplement: Iron Folic Acid Supplement — Standard of Care Intervention
  Arms: IFA + Standard of Care

SUMMARY:
The aim of this implementation research is to compare how different implementation strategies influence the acceptability and adherence to antenatal supplement use in pregnancy.

DETAILED DESCRIPTION:
In the past several decades, the République du Mali (Mali) has achieved reductions in both maternal mortality ratio and neonatal mortality rate. However, with an estimated 562 maternal deaths per 100,000 live births and 65.8 infant deaths per 1,000 births, substantial changes to maternal child health services will likely need to be implemented to realize the benefits of universal healthcare for mothers and children and recover from the damaging impacts of colonialism and conflict. The prevalence of low birth weight (<2.5 kg) among children whose birth weights are known is estimated to be approximately 16%, but is likely underestimated. The Malian decentralized health system places antenatal care (ANC) at Centre de Santé Communautaire (CSCOM), a type of community-based health center. Approximately 36% of women in Mali access ANC in the first trimester. Within the context of ANC, the current national policy in Mali recommends that pregnant women take daily IFA supplements that contain 60 mg of iron and 400 μg of folic acid starting at the first ANC contact and ending three months after delivery. However, recent DHS data indicates that coverage of iron for pregnant women for at least 90 days has remained sub-optimal, and may be decreasing, with only 28% of women taking iron tablets for at least 90 days during their last pregnancy.

While IFA supplements have been a component of the "gold standard" of antenatal nutritional care for decades, there is clear and consistent evidence from clinical trials that MMS provide additional benefits over IFA in reducing adverse pregnancy outcomes. As compared to IFA, MMS performs better in reducing the occurrence of small for gestational age (SGA), low birth weight (LBW), preterm birth, and stillbirth. MMS performs even better than IFA with respect to pregnancy outcomes and infant survival when used by pregnant women who are anemic or underweight. Further, MMS has been demonstrated to be safe, cost-effective, and possible to produce at price parity with IFA. In 2020, the WHO released updated ANC guidelines recommending the use of MMS containing iron and folic acid in the context of rigorous research, including implementation research (IR) to establish the impact of switching from IFA supplements to MMS, including evaluation of uptake, acceptability, adherence, and cost-effectiveness.

This implementation research study design will facilitate answering the following questions, all of which were deemed to be of importance when considering the potential switch from supplementation with iron and folic acid (IFA) to multiple micronutrient supplementation (MMS) in the Malian context:

1. How does adherence to antenatal supplement use compare across study arms?
2. How does acceptability of antenatal supplements compare across study arms for both ANC clients and midwives?
3. What level of acceptability is associated with a novel counseling package for MMS?
4. What is the cost-effectiveness of switching from IFA to MMS in the Malian context?

ELIGIBILITY:
INCLUSION CRITERIA:

Sample Group 1: Pregnant Women

Potential supplementation trial participants must meet all the following criteria to be eligible for inclusion in the study:

1. Age 18 years or older at screening.
2. At time of enrollment, able and willing to comply with all study requirements and complete all study procedures.
3. Able and willing to provide verbal informed consent to be screened for and to take part in the study.
4. Intention to stay within study catchment area for study duration and willingness to give adequate locator information, as defined in site standard operating procedures (SOPs).
5. Presenting for first ANC visit.
6. Pregnant, as confirmed by at least one of the following:

   1. Uterine examination
   2. Urine human chorionic gonadotropin (HCG)
   3. Ultrasound

Sample Group 2: Midwives

Midwives who participated in delivery of the intervention will be recruited from the six health center study sites. Inclusion criteria includes the provision of verbal informed consent.

Sample Group 3: Pharmacists

Pharmacists who participated in delivery of the intervention will be recruited from the six health center study sites. Inclusion criteria includes the provision of verbal informed consent.

Sample Group 4: Family Members

Family members (e.g., male partners and mothers/mothers-in-law) will be recruited based on participation of their female family member in the study protocol. Inclusion criteria includes the provision of verbal informed consent.

EXCLUSION CRITERIA:

Sample Group 1: Pregnant Women

Potential supplementation trial participants who meet any of the following criteria will be excluded from the study:

1. At time of enrollment, evidence of gestational age greater than 26 0/7 weeks, using one or more of the following methods: a) Uterine examination, b) First day of last normal menstrual period, and c) Ultrasound
2. As determined by the site investigator, any significant uncontrolled active or chronic cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, respiratory, immunologic disorder, or infectious disease. Note: examples of uncontrolled conditions include but are not limited to the following: HIV not virally suppressed, COVID-19 infection, symptomatic malaria infection.
3. Has any other condition that, in the opinion of the site investigator, would preclude verbal informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.
4. At time of enrollment, any known condition requiring routine antenatal care to take place at a location other than the study site CSCOM, e.g., Rh- negative status.
5. At enrollment, reports either of the following: a) Participation in any research study involving drugs, vaccines, or medical devices during the current pregnancy, b) Expected to participate in other research studies involving drugs, vaccines, or medical devices for the duration of study participation

Sample Group 2: Midwives

Potential participants who do not provide verbal informed consent will not be included.

Sample Group 3: Pharmacists

Potential participants who do not provide verbal informed consent will not be included.

Sample Group 4: Family Members

Potential participants who do not provide verbal informed consent will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 486 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Adherence to the Antenatal Supplement Intervention (pill count) | 4 weeks post-enrollment (ANC-2)
  Adherence assessment (pill count report)
Adherence to the Antenatal Supplement Intervention (pill count) | ANC follow-up visit (ANC-3) - approximately 4-6 weeks after ANC-2
  Adherence assessment (pill count report)
Adherence to the Antenatal Supplement Intervention (pill count) | ANC follow-up visit (ANC-4) - approximately 4-6 weeks after ANC-3
  Adherence assessment (pill count report)
Adherence to the Antenatal Supplement Intervention (pill count) | ANC follow-up visit (ANC-5) - approximately 4-6 weeks after ANC-4
  Adherence assessment (pill count report)
Adherence to the Antenatal Supplement Intervention (pill count) | ANC follow-up visit (ANC-6) - approximately 4-6 weeks after ANC-5
  Adherence assessment (pill count report)
Adherence to the Antenatal Supplement Intervention (pill count) | ANC follow-up visit (ANC-7) - approximately 4-6 weeks after ANC-6
  Adherence assessment (pill count report)
Adherence to the Antenatal Supplement Intervention (pill count) | ANC follow-up visit (ANC-8) - approximately 4-6 weeks after ANC-7
  Adherence assessment (pill count report)
Adherence to the Antenatal Supplement Intervention (pill count) | Postnatal visit (6 weeks after delivery of infant)
  Adherence assessment (pill count report)
Adherence to Antenatal Supplement Intervention (self report) | 4 weeks post-enrollment (ANC-2)
  Interviewer administered retrospective self report
Adherence to Antenatal Supplement Intervention (self report) | ANC follow-up visit (ANC-3) - approximately 4-6 weeks after ANC-2
  Interviewer administered retrospective self report
Adherence to Antenatal Supplement Intervention (self report) | ANC follow-up visit (ANC-4) - approximately 4-6 weeks after ANC-3
  Interviewer administered retrospective self report
Adherence to Antenatal Supplement Intervention (self report) | ANC follow-up visit (ANC-5) - approximately 4-6 weeks after ANC-4
  Interviewer administered retrospective self report
Adherence to Antenatal Supplement Intervention (self report) | ANC follow-up visit (ANC-6) - approximately 4-6 weeks after ANC-5
  Interviewer administered retrospective self report
Adherence to Antenatal Supplement Intervention (self report) | ANC follow-up visit (ANC-7) - approximately 4-6 weeks after ANC-6
  Interviewer administered retrospective self report
Adherence to Antenatal Supplement Intervention (self report) | ANC follow-up visit (ANC-8) - approximately 4-6 weeks after ANC-7
  Interviewer administered retrospective self report
Adherence to Antenatal Supplement Intervention (self report) | Postnatal visit (6 weeks after delivery of infant)
  Interviewer administered retrospective self report

SECONDARY OUTCOMES:
Acceptability of Antenatal Supplement (i.e., pregnant women) | At 4 weeks post-enrollment (ANC-2)
  Proportion of ANC clients (i.e., pregnant women) who find the antenatal supplement to be acceptable.
Acceptability of Antenatal Supplement (i.e., pregnant women) | ANC follow-up visit (ANC-3) - approximately 4-6 weeks after ANC-2
  Proportion of ANC clients (i.e., pregnant women) who find the antenatal supplement to be acceptable.
Acceptability of Antenatal Supplement (i.e., pregnant women) | ANC follow-up visit (ANC-4) - approximately 4-6 weeks after ANC-3
  Proportion of ANC clients (i.e., pregnant women) who find the antenatal supplement to be acceptable.
Acceptability of Antenatal Supplement (i.e., pregnant women) | ANC follow-up visit (ANC-5) - approximately 4-6 weeks after ANC-4
  Proportion of ANC clients (i.e., pregnant women) who find the antenatal supplement to be acceptable.
Acceptability of Antenatal Supplement (i.e., pregnant women) | ANC follow-up visit (ANC-6) - approximately 4-6 weeks after ANC-5
  Proportion of ANC clients (i.e., pregnant women) who find the antenatal supplement to be acceptable.
Acceptability of Antenatal Supplement (i.e., pregnant women) | ANC follow-up visit (ANC-7) - approximately 4-6 weeks after ANC-6
  Proportion of ANC clients (i.e., pregnant women) who find the antenatal supplement to be acceptable.
Acceptability of Antenatal Supplement (i.e., pregnant women) | ANC follow-up visit (ANC-8) - approximately 4-6 weeks after ANC-7
  Proportion of ANC clients (i.e., pregnant women) who find the antenatal supplement to be acceptable.
Acceptability of Antenatal Supplement (i.e., pregnant women) | Postnatal visit (6 weeks after delivery of infant)
  Proportion of ANC clients (i.e., pregnant women) who find the antenatal supplement to be acceptable.
Acceptability of Antenatal Counseling (i.e., pregnant women) | At 4 weeks post-enrollment (ANC-2)
  Proportion of ANC clients (i.e., pregnant women) who find the antenatal counseling to be acceptable.
Acceptability of Antenatal Counseling (i.e., pregnant women) | ANC follow-up visit (ANC-3) - approximately 4-6 weeks after ANC-2
  Proportion of ANC clients (i.e., pregnant women) who find the antenatal counseling to be acceptable. Perceptions of midwives, pharmacists, and family members on counseling acceptability.
Acceptability of Antenatal Counseling (i.e., pregnant women) | ANC follow-up visit (ANC-4) - approximately 4-6 weeks after ANC-3
  Proportion of ANC clients (i.e., pregnant women) who find the antenatal counseling to be acceptable. Perceptions of midwives, pharmacists, and family members on counseling acceptability.
Acceptability of Antenatal Counseling (i.e., pregnant women) | ANC follow-up visit (ANC-5) - approximately 4-6 weeks after ANC-4
  Proportion of ANC clients (i.e., pregnant women) who find the antenatal counseling to be acceptable. Perceptions of midwives, pharmacists, and family members on counseling acceptability.
Acceptability of Antenatal Counseling (i.e., pregnant women) | ANC follow-up visit (ANC-6) - approximately 4-6 weeks after ANC-5
  Proportion of ANC clients (i.e., pregnant women) who find the antenatal counseling to be acceptable. Perceptions of midwives, pharmacists, and family members on counseling acceptability.
Acceptability of Antenatal Counseling (i.e., pregnant women) | ANC follow-up visit (ANC-7) - approximately 4-6 weeks after ANC-6
  Proportion of ANC clients (i.e., pregnant women) who find the antenatal counseling to be acceptable. Perceptions of midwives, pharmacists, and family members on counseling acceptability.
Acceptability of Antenatal Counseling (i.e., pregnant women) | ANC follow-up visit (ANC-8) - approximately 4-6 weeks after ANC-7
  Proportion of ANC clients (i.e., pregnant women) who find the antenatal counseling to be acceptable. Perceptions of midwives, pharmacists, and family members on counseling acceptability.
Acceptability of Antenatal Counseling (i.e., pregnant women) | Postnatal visit (6 weeks after delivery of infant)
  Proportion of ANC clients (i.e., pregnant women) who find the antenatal counseling to be acceptable.
Acceptability of Antenatal Supplement (i.e., midwives) - Global Acceptability Assessment Form (supplement) and Focus Group Discussion Guide | Within 2 months of study completion
  Proportion of midwives who find the antenatal supplement to be acceptable.
Acceptability of Antenatal Supplement (i.e., pharmacists) - Global Acceptability Assessment Form (supplement) and Focus Group Discussion Guide | Within 2 months of study completion
  Proportion of pharmacists who find the antenatal supplement to be acceptable.
Acceptability of Antenatal Supplement (i.e., family members) - Global Acceptability Assessment Form (supplement) and Focus Group Discussion Guide | Within 2 months of study completion
  Proportion of family members of ANC clients who find the antenatal supplement to be acceptable.
Acceptability of Antenatal Counseling (i.e., midwives) - Global Acceptability Assessment Form (counseling) and Focus Group Discussion Guide | Within 2 months of study completion
  Proportion of midwives who find the antenatal counseling to be acceptable.
Acceptability of Antenatal Counseling (i.e., pharmacists) - Global Acceptability Assessment Form (counseling) and Focus Group Discussion Guide | Within 2 months of study completion
  Proportion of pharmacists who find the antenatal counseling to be acceptable.
Acceptability of Antenatal Counseling (i.e., family members) - Global Acceptability Assessment Form (counseling) and Focus Group Discussion Guide | Within 2 months of study completion
  Proportion of family members of ANC clients who find the antenatal counseling to be acceptable.

OTHER OUTCOMES:
Pregnancy Outcome - Maternal Hemoglobin (Exploratory outcomes) | Collected at delivery via health record review
  Maternal hemoglobin collected at delivery admission as reported on health record.
Pregnancy Outcome - Gestational Age (Exploratory outcomes) | Collected at delivery via health record review
  Gestational age collected at delivery as reported on health record (best obstetric estimate)
Birth outcome (Exploratory outcomes) | Collected at delivery via health record review
  Birthweight as reported on health record.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen M Hurley, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Lisa Noguchi, PhD, Study Director — Jhpiego; Samba Sow, MD, Study Director — Center for Vaccine Development - Mali
Locations (1):
- JPIEGO Mali, Bamako, Mali

IPD SHARING:
Plan to Share IPD: Yes
After data collection and analysis, Johns Hopkins Biostatistics Center (JHBC) and Johns Hopkins University (JHU) investigators will de-identify the data. The de-identified data will be shared with Research Triangle Institute (RTI) who is responsible for managing access to the shared data from all partners across the Gates ANC-PNC research collaborative, of which Jhpiego is a partner. This data will be collected and stored through the Synapse platform. The data will not be individually identifiable. The investigators will also adhere to JHBC's data sharing policies.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After data collection and analysis. The individual personal data (IPD) will be share after the data analysis for the described research questions (see above) is complete
Access Criteria: The data will be collected and stored through the Synapse platform. The data will not be individually identifiable. Investigators will also adhere to JHBC's data sharing policies.

REFERENCES:
- [Background] Bourassa MW, Osendarp SJM, Adu-Afarwuah S, Ahmed S, Ajello C, Bergeron G, Black R, Christian P, Cousens S, de Pee S, Dewey KG, Arifeen SE, Engle-Stone R, Fleet A, Gernand AD, Hoddinott J, Klemm R, Kraemer K, Kupka R, McLean E, Moore SE, Neufeld LM, Persson LA, Rasmussen KM, Shankar AH, Smith E, Sudfeld CR, Udomkesmalee E, Vosti SA. Review of the evidence regarding the use of antenatal multiple micronutrient supplementation in low- and middle-income countries. Ann N Y Acad Sci. 2019 May;1444(1):6-21. doi: 10.1111/nyas.14121. Epub 2019 May 27. PMID 31134643
- [Background] Engle-Stone R, Kumordzie SM, Meinzen-Dick L, Vosti SA. Replacing iron-folic acid with multiple micronutrient supplements among pregnant women in Bangladesh and Burkina Faso: costs, impacts, and cost-effectiveness. Ann N Y Acad Sci. 2019 May;1444(1):35-51. doi: 10.1111/nyas.14132. Epub 2019 May 27. PMID 31134641
- [Background] Demographic Health Survey Mali 2018. https://link.edgepilot.com/s/58ae5387/4L1KP3pdmU6VyyFqGxSdsQ?u=https://dhsprogram.com/methodology/survey/survey-display-517.cfm
- [Background] Institut National de la Statistique - INSTAT, Cellule de Planification et de Statistique Secteur Santé-Développement Social et Promotion de la Famille CPS/SS-DS-PF et ICF. 2019. Enquête Démographique et de Santé au Mali 2018.Bamako, Mali et Rockville, Maryland, USA : INSTAT, CPS/SS-DS-PF et ICF.
- [Background] Keats EC, Haider BA, Tam E, Bhutta ZA. Multiple-micronutrient supplementation for women during pregnancy. Cochrane Database Syst Rev. 2019 Mar 14;3(3):CD004905. doi: 10.1002/14651858.CD004905.pub6. PMID 30873598
- [Background] Smith ER, Shankar AH, Wu LS, Aboud S, Adu-Afarwuah S, Ali H, Agustina R, Arifeen S, Ashorn P, Bhutta ZA, Christian P, Devakumar D, Dewey KG, Friis H, Gomo E, Gupta P, Kaestel P, Kolsteren P, Lanou H, Maleta K, Mamadoultaibou A, Msamanga G, Osrin D, Persson LA, Ramakrishnan U, Rivera JA, Rizvi A, Sachdev HPS, Urassa W, West KP Jr, Zagre N, Zeng L, Zhu Z, Fawzi WW, Sudfeld CR. Modifiers of the effect of maternal multiple micronutrient supplementation on stillbirth, birth outcomes, and infant mortality: a meta-analysis of individual patient data from 17 randomised trials in low-income and middle-income countries. Lancet Glob Health. 2017 Nov;5(11):e1090-e1100. doi: 10.1016/S2214-109X(17)30371-6. PMID 29025632
- [Background] WHO antenatal care recommendations for a positive pregnancy experience: Nutritional interventions update: Multiple micronutrient supplements during pregnancy [Internet]. Geneva: World Health Organization; 2020. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK560384/ PMID 32783435
- [Background] United Nations Interagency Group for Child Mortality Estimation. Level and trend in child mortality report. 2017
- [Background] Alkema L, Chou D, Hogan D, Zhang S, Moller AB, Gemmill A, Fat DM, Boerma T, Temmerman M, Mathers C, Say L; United Nations Maternal Mortality Estimation Inter-Agency Group collaborators and technical advisory group. Global, regional, and national levels and trends in maternal mortality between 1990 and 2015, with scenario-based projections to 2030: a systematic analysis by the UN Maternal Mortality Estimation Inter-Agency Group. Lancet. 2016 Jan 30;387(10017):462-74. doi: 10.1016/S0140-6736(15)00838-7. Epub 2015 Nov 13. PMID 26584737